CLINICAL TRIAL: NCT03317002
Title: A 12-week, Randomized, Single-blind, Placebo-controlled, Multi-centre, Parallel Group, Phase IIa Study to Evaluate Efficacy, Safety and Tolerability of Oral AZD5718 After 4 and 12-weeks of Treatment in Patients With Coronary Artery Disease (CAD)
Brief Title: AZD5718 Phase IIa Study to Evaluate Efficacy, Safety and Tolerability of Oral AZD5718 in Patients With Coronary Artery Disease (CAD).
Acronym: FLAVOUR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D7550C00003
Record Dates: First submitted 2017-10-05; First posted 2017-10-23 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — AZD5718

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AZD5718 Dose A (Experimental): AZD5718 Dose A once daily
  Interventions: Drug: AZD5718
- AZD5718 Dose B (Experimental): AZD5718 Dose B once daily
  Interventions: Drug: AZD5718
- Placebo (Placebo Comparator): Matching placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5718 — Oral dose of AZD5718 (tablet)
  Arms: AZD5718 Dose A
Drug: AZD5718 — Oral dose of AZD5718 (tablet)
  Arms: AZD5718 Dose B
Drug: Placebo — Matching placebo (tablet)
  Arms: Placebo

SUMMARY:
This is a randomized, single-blind, placebo-controlled, parallel-group, multicentre study in patients with CAD. The study will be conducted at approximately 10 centres in 3 countries. Approximately 138 CAD patients will be randomized to AZD5718 or placebo (treatment duration 12 weeks).

DETAILED DESCRIPTION:
This is a randomized, single-blind, placebo-controlled, parallel-group, multicentre study in patients with CAD. The study will be conducted at approximately 10 centres in 3 countries (Denmark, Finland and Sweden).

Patients suitable for the study will be identified and screened for eligibility after being hospitalized for Acute Coronary Syndrome (ACS) (Visit 1) comprising ST Elevation Myocardial Infarction (STEMI) or Non-ST Elevation Myocardial Infarction (non-STEMI). At Visit 1, after signing informed consent, study measurements will take place at days 1, 2, 3 and 5 post ACS, where feasible. It is planned that approximately 138 CAD patients will be randomized to ensure at least 66 evaluable patients receiving AZD5718 Dose B or placebo are included with 12 weeks treatment. For supporting dose selection in future studies, a treatment arm with 28 randomized patients receiving AZD5718 Dose A is included in the study. The study was originally designed to be a 4-week study and was amended to be a 12-week study. Therefore, the total number of patients is greater than required for a 12 weeks study (about 100), since some patients will only have 4 weeks of treatment.

An evaluable patient is defined as a patient with a valid Coronary Flow Velocity Reserve (CFVR) measurement at Visit 2 and one post baseline visit as judged by the CFVR Core lab.

On Day 1 (Visit 2), 7 to 28 days after the ACS event, patients willing to participate in the study will complete the screening procedure and, if eligible, be randomized. Treatment duration will be 12 weeks. During the treatment phase, patients will come in to the clinic for study measurements at 2 weeks (visit 3), 4 weeks (visit 4), 8 weeks (visit 4b) and 12 weeks (visit 4c).

A follow-up visit (Visit 5) will be performed at 4 weeks (±4 days) after last dose in order to ensure safety and well-being of the patients

ELIGIBILITY:
Inclusion Criteria:

* Males and females of non-childbearing potential
* Age ≥18 to ≤75
* Body Mass Index (BMI) ≥18 to ≤35 kg/m2
* CAD patients, here defined as:

ACS 7-28 days prior to study randomization (ACS defined as STEMI, non STEMI event documented by Electrocardiogram (ECG), cardiac enzymes [troponin] and angiogram) Provision of signed and dated, written informed consent prior to any study specific procedures

Exclusion Criteria:

* Uncontrolled Type 1 or Type 2 diabetes defined as haemoglobin A1c (HbA1c) Diabetes
* Control and Complications Trial (DCCT)> 9% or International Federation of Clinical Chemistry (IFCC) >74.9 mmol/mol
* Patients with atrial fibrillation (chronic or current) or history of ventricular tachycardia requiring therapy for termination, or symptomatic sustained ventricular tachycardia or sick sinus syndrome or Atrioventricular blockage degree 2-3
* Prior coronary artery by-pass graft (Coronary artery bypass grafting) to Left Anterior Descending artery (LAD)
* Left ventricle ejection fraction < 30%
* Unacceptable level of angina despite maximal medical therapy or unstable angina at entry
* Canadian Cardiovascular Society (CCS) ≥ 3 (Visit 1 or Visit 2)
* Stroke within the previous 6 months from ACS or ongoing treatment with Persantin or Asasantin
* Chronic use of anticoagulants on therapeutic dose (not including thrombosis prophylaxis) during the study
* Planned additional cardiac intervention (e.g., Percutaneous coronary intervention (PCI), Coronary artery bypass grafting (CABG) within next 6 months
* New York Heart Association (NYHA) class III-IV heart failure or decompensated heart failure at discharge or hospitalization for exacerbation of chronic heart failure within the previous 3 months from ACS
* Previously known severe renal disease (Chronic Kidney Disease (CKD) stage 4 or 5) or previously known creatinine clearance calculated by Cockcroft Gault equation <30 ml/min*m2
* Known allergy to adenosine and mannitol, or experience of previous adverse effects of adenosine stress testing.
* Participation in another interventional clinical study with an investigational pharmaceutical product during the last 3 months also including drug eluting stents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- Denmark (3):
  - Research Site, Aarhus
  - Research Site, Frederiksberg
  - Research Site, Odense C
- Finland (2):
  - Research Site, Kuopio
  - Research Site, Turku
- Sweden (4):
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Stockholm
  - Research Site, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Prescott E, Angeras O, Erlinge D, Grove EL, Hedman M, Jensen LO, Pernow J, Saraste A, Akerblom A, Svedlund S, Rudvik A, Knochel J, Lindstedt EL, Garkaviy P, Gan LM, Gabrielsen A. Safety and efficacy of the 5-lipoxygenase-activating protein inhibitor AZD5718 in patients with recent myocardial infarction: The phase 2a FLAVOUR study. Int J Cardiol. 2022 Oct 15;365:34-40. doi: 10.1016/j.ijcard.2022.07.016. Epub 2022 Jul 14. PMID 35842004
- See also: redacted Statistical Analysis Plan — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7550C00003&attachmentIdentifier=bfc8ef9d-0ec7-4ad9-9153-27fb6e2d880e&fileName=Statistical_Analysis_Plan_redacted.pdf&versionIdentifier=
- See also: redacted Clinical Study Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7550C00003&attachmentIdentifier=72c1cf18-0bad-4d45-a0cd-640350986d43&fileName=Clinical_Study_Protocol_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 3 countries at 9 sites; 3 in Denmark, 2 in Finland and 4 in Sweden.
Pre-assignment Details: Participants underwent a screening visit between 2 and within 27 days before receiving the first dose of IP.
Groups:
- AZD5718 (200 mg): AZD5718 (200 mg)
- AZD5718 (50 mg): AZD5718 (50 mg)
- Placebo: Placebo
Period: Overall Study
Arm/Group | AZD5718 (200 mg) | AZD5718 (50 mg) | Placebo
Started | 52 | 25 | 52
Completed | 50 | 24 | 51
Not Completed | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD5718 (200 mg) | AZD5718 (50 mg) | Placebo | Total
Number analyzed (Participants) | 52 | 25 | 51 | 128
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (8.21) | 61.4 (8.12) | 61.1 (8.51) | 61.5 (8.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 10 | 17
  Male | 45 | 25 | 41 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 51 | 25 | 51 | 127
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 52 | 25 | 50 | 127
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Creatinine-normalized u-LTE4 at Week 4
Description: Creatinine-normalized u-LTE4 is calculated as uLTE4/creatinine
Time Frame: Baseline and 4 weeks
Population: Number of participants analysed differs from participant flow module due to missing data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | AZD5718 (200 mg) | AZD5718 (50 mg) | Placebo
Number analyzed (Participants) | 49 | 24 | 50
Ratio | 0.04 (92.55) | 0.09 (84.32) | 1.09 (44.38)
Statistical Analysis 1: Comparison: AZD5718 (200 mg) vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Ratio = 0.04, 95% CI 1-sided [upper limit 0.05]
Statistical Analysis 2: Comparison: AZD5718 (50 mg) vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis; Ratio = 0.08, 95% CI 1-sided [upper limit 0.10]

2. Secondary Outcome: Change From Baseline in Creatinine-normalized u-LTE4 at Week 12
Description: Creatinine-normalized u-LTE4 is calculated as uLTE4/creatinine
Time Frame: Baseline and 12 weeks
Population: Number of participants analysed differs from participant flow module due to missing data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | AZD5718 (200 mg) | AZD5718 (50 mg) | Placebo
Number analyzed (Participants) | 29 | 18 | 36
Ratio | 0.04 (92.55) | 0.09 (84.32) | 1.09 (44.38)
Statistical Analysis 1: Comparison: AZD5718 (200 mg) vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Ratio = 0.04, 95% CI 1-sided [upper limit 0.05]
Statistical Analysis 2: Comparison: AZD5718 (50 mg) vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis; Ratio = 0.09, 95% CI 1-sided [upper limit 0.12]

3. Secondary Outcome: Change From Baseline in CFVR at Week 12
Description: CFVR = Coronary Flow Velocity Reserve = LAD(hyperaemic)/LAD(rest)
Time Frame: Baseline and 12 weeks
Population: Number of participants analysed differs from participant flow module due to missing data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | AZD5718 (200 mg) | AZD5718 (50 mg) | Placebo
Number analyzed (Participants) | 16 | 11 | 24
Ratio | 0.93 (23.64) | 0.98 (39.53) | 1.16 (33.46)

4. Secondary Outcome: Change From Baseline in CFVR at Week 4
Description: CFVR = Coronary Flow Velocity Reserve = LAD(hyperaemic)/LAD(rest)
Time Frame: Baseline and 4 weeks
Population: Number of participants analysed differs from participant flow module due to missing data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | AZD5718 (200 mg) | AZD5718 (50 mg) | Placebo
Number analyzed (Participants) | 36 | 16 | 38
Ratio | 1.03 (28.34) | 1.15 (31.47) | 1.08 (33.16)

5. Secondary Outcome: Summary of Plasma Concentrations of AZD5718
Time Frame: 16 weeks
Population: Number of participants analysed differs from participant flow module due to missing data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | AZD5718 (200 mg) | AZD5718 (50 mg)
Number analyzed (Participants) | 52 | 25
nmol/L
  Baseline: 1-8 Hours Post-Dose | 611.88 (234.50) | 47.88 (497.86)
  2 weeks (Visit 3): 20-28 Hours Post-Dose | 59.36 (90.97) | 16.57 (127.80)
  4 weeks (Visit 4): Pre-Dose | 48.00 (68.17) | 11.01 (60.70)
  4 weeks (Visit 4): 0-2 Hours Post-Dose | 339.28 (243.04) | 38.68 (159.56)
  4 weeks (Visit 4): 2-4 Hours Post-Dose | 919.22 (51.26) | 148.64 (71.86)
  4 weeks (Visit 4): 4-8 Hours Post-Dose | 649.09 (49.89) | 105.40 (52.16)
  12 weeks (Visit 4c): Pre-Dose | 65.39 (91.52) | 13.97 (88.12)
  16 weeks (Visit 5) - FUP 1 month | 0.51 (16.39) | 0.50 (0.00)

6. Secondary Outcome: Change From Baseline in LAD Hypereamic Flow at 4 Weeks
Description: LAD=Left Anterior Descending
Time Frame: Baseline and 4 weeks
Population: Number of participants analysed differs from participant flow module due to missing data
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | AZD5718 (200 mg) | AZD5718 (50 mg) | Placebo
Number analyzed (Participants) | 36 | 16 | 38
m/sec | 0.02 (0.16) | 0.04 (0.16) | 0.03 (0.17)

7. Secondary Outcome: Change From Baseline in LVEF at 4 Weeks
Description: LVEF=Left Ventricular Ejection Fraction
Time Frame: Baseline and 4 weeks
Population: Number of participants analysed differs from participant flow module due to missing data
Measure: Mean (Standard Deviation); unit: percent LVEF
Arm/Group | AZD5718 (200 mg) | AZD5718 (50 mg) | Placebo
Number analyzed (Participants) | 46 | 22 | 45
percent LVEF | -0.23 (5.30) | 2.70 (6.39) | 0.48 (5.00)

8. Secondary Outcome: Change From Baseline in LV Longitudinal Early Diastolic Strain Rate at 4 Weeks
Description: LV=Left Ventricular
Time Frame: Baseline and 4 weeks
Population: Number of participants analysed differs from participant flow module due to missing data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/s
Arm/Group | AZD5718 (200 mg) | AZD5718 (50 mg) | Placebo
Number analyzed (Participants) | 43 | 19 | 44
1/s | 1.02 (30.61) | 0.98 (33.55) | 1.03 (30.45)

9. Secondary Outcome: Change From Baseline in LV-GLS at Rest at Week 4
Description: LV-GLS = Left Ventricular Global Longitudinal Strain
Time Frame: Baseline and 4 weeks
Population: Number of participants analysed differs from participant flow module due to missing data
Measure: Mean (Standard Deviation); unit: Percent LV-GLS
Arm/Group | AZD5718 (200 mg) | AZD5718 (50 mg) | Placebo
Number analyzed (Participants) | 43 | 17 | 42
Percent LV-GLS | -0.41 (3.00) | 0.34 (2.47) | -0.63 (2.61)

10. Secondary Outcome: Change From Baseline in LV-GCS at Rest at Week 4
Description: LV-GCS = Left Ventricular Global Circumferential Strain
Time Frame: Baseline and 4 weeks
Population: Number of participants analysed differs from participant flow module due to missing data
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | AZD5718 (200 mg) | AZD5718 (50 mg) | Placebo
Number analyzed (Participants) | 39 | 16 | 34
Percent | 0.34 (7.24) | 1.71 (5.40) | -1.88 (6.78)

11. Secondary Outcome: Change From Baseline in LAD Resting Mean Diastolic Flow Velocity at 4 Weeks
Description: LAD=Left Anterior Descending
Time Frame: Baseline and 4 weeks
Population: Number of participants analysed differs from participant flow module due to missing data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: m/sec
Arm/Group | AZD5718 (200 mg) | AZD5718 (50 mg) | Placebo
Number analyzed (Participants) | 36 | 16 | 38
m/sec | 1.01 (23.31) | 0.92 (23.68) | 0.99 (20.14)

ADVERSE EVENTS:
Time Frame: Treatment period, up to 12 weeks
Arm/Group | AZD5718 (200 mg) | AZD5718 (50 mg) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/25 | 0/51
Serious Adverse Events (participants affected / at risk) | 4/52 | 3/25 | 4/51
Other Adverse Events (participants affected / at risk) | 27/52 | 12/25 | 22/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD5718 (200 mg) (N=52) | AZD5718 (50 mg) (N=25) | Placebo (N=51)
Post procedural sepsis (Infections and infestations) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chest pain (General disorders) | 2 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 0.03% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD5718 (200 mg) (N=52) | AZD5718 (50 mg) (N=25) | Placebo (N=51)
Nasopharyngitis (Infections and infestations) | 6 | 4 | 7
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1
Dizziness (Nervous system disorders) | 5 | 2 | 4
Headache (Nervous system disorders) | 1 | 1 | 2
Chest pain (General disorders) | 3 | 1 | 3
Fatigue (General disorders) | 3 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 4
Alanine aminotransferase increased (Investigations) | 0 | 0 | 4
Anxiety (Psychiatric disorders) | 2 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT03317002/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/02/NCT03317002/SAP_001.pdf